CLINICAL TRIAL: NCT00854334
Title: Co-existent OSA and Obesity: Finding NEAT Targets for Intervention
Brief Title: Co-existent Obstructive Sleep Apnea (OSA) and Obesity: Finding Non-exercise Activity Thermogenesis (NEAT) Targets for Intervention
Status: Completed | Type: Observational
Sponsor: Katz, Sherri Lynne, M.D. (Individual)
Responsible Party: Principal Investigator, Dr. Sherry Lynn Katz, Katz, Sherri Lynne, M.D., Children's Hospital of Eastern Ontario
Other Study IDs: Neat-OSA-001
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Childhood Obesity; Childhood Obstructive Sleep Apnea
Keywords: Sleep; Overweight; Physical activity; Appetite; NEAT
MeSH Terms: conditions — Pediatric Obesity; Overweight; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1.: Children with both obesity and obstructive sleep apnea
- 2: Children without the presence of both obesity and obstructive sleep apnea

SUMMARY:
Rationale: Obesity is an increasing childhood epidemic in Canada. Obstructive sleep apnea (OSA) is a complication of obesity which causes cardiovascular disease, reduced quality of life, and premature death. While the complex interactions between obesity and OSA are not entirely clear, we hypothesize that these conditions may compound each other by:

1. decreasing physical activity and total energy expenditure by reducing both non-exercise physical pursuits (NEAT- non-exercise activity thermogenesis) and purposeful physical activity.
2. alterations in the secretion of appetite-controlling hormones, which may lead to increases in energy intake.

Objective: To determine whether the presence of both obesity and OSA in children is associated with a decrease in physical activity and alterations in appetite-regulating hormones greater than those seen in either condition alone or compared to controls.

Methods: Comparison of children 10-17 years with obesity and OSA, obesity alone, OSA alone and neither condition, for the following outcomes: (1) NEAT (kcal/day) (2) Physical activity behavior, appetite regulating hormone profile and self-report appetite assessment.

Unique Aspects: This study combines expertise in sleep medicine, exercise physiology and obesity. Conclusions from this study will better characterize this high-risk clinical population so that innovative strategies targeting improvements in lifestyle behaviors can be developed.

ELIGIBILITY:
Inclusion Criteria:

* age 10-17 years
* coming for polysomnography at the Children's Hospital of Eastern Ontario

Exclusion Criteria:

* children receiving treatment for OSA with CPAP (continuous positive airway pressure) or bi-level therapy
* craniofacial abnormalities
* genetic syndromes
* neuromuscular disease
* tracheostomy
* medications that may affect appetite or energy balance (systemic corticosteroids)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited from those scheduled to undergo polysomnography in the sleep laboratory at the Children's Hospital of Eastern Ontario
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
NEAT (kcal/day) | 10 day period

SECONDARY OUTCOMES:
Physical activity behavior (minutes of moderate-vigorous physical activity as directly measured by accelerometry), appetite regulating hormone profile and self-report appetite assessment. | 10 day period

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital of Eastern Ontario, Ottawa, Ontario, Canada